CLINICAL TRIAL: NCT05644301
Title: INflammation-based Stratification for Immune-Targeted Augmentation in Major Depressive
Brief Title: INflammation-based Stratification for Immune-Targeted Augmentation in Major Depressive Disorder
Acronym: INSTA-MD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Research Foundation Flanders (Other); KU Leuven (Other); Vrije Universiteit Brussel (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Manuel Morrens, Professor Doctor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T001222N
Record Dates: First submitted 2022-11-24; First posted 2022-12-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; Inflammation
Keywords: Immunopsychiatry; Celecoxib; Minocyclin; Inflammation; Randomised Controlled Clinical Trial
MeSH Terms: conditions — Depressive Disorder, Major; Inflammation; cyclopia sequence | interventions — Celecoxib; Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- High Sensitive C-reactive Protein (hs-CRP) < 3mg/L: Minocyclin + Treatment As Usual (TAU) (Active Comparator)
  Interventions: Drug: Minocyclin
- High Sensitive C-reactive Protein (hs-CRP) < 3mg/L: Celecoxib + Treatment As Usual (TAU) (Active Comparator)
  Interventions: Drug: Celecoxib
- High Sensitive C-reactive Protein (hs-CRP) < 3mg/L: Placebo + Treatment As Usual (TAU) (Placebo Comparator)
  Interventions: Drug: Placebo
- High Sensitive C-reactive Protein (hs-CRP) > 3mg/L: Minocyclin + Treatment As Usual (TAU) (Active Comparator)
  Interventions: Drug: Minocyclin
- High Sensitive C-reactive Protein (hs-CRP) > 3mg/L: Celecoxib + Treatment As Usual (TAU) (Active Comparator)
  Interventions: Drug: Celecoxib
- High Sensitive C-reactive Protein (hs-CRP) > 3mg/L: Placebo + Treatment As Usual (TAU) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Oral capsule, 200 mg, twice daily, for 12 weeks
  Arms: High Sensitive C-reactive Protein (hs-CRP) < 3mg/L: Celecoxib + Treatment As Usual (TAU); High Sensitive C-reactive Protein (hs-CRP) > 3mg/L: Celecoxib + Treatment As Usual (TAU)
Drug: Minocyclin — Oral capsule, 100 mg, twice daily, for 12 weeks
  Arms: High Sensitive C-reactive Protein (hs-CRP) < 3mg/L: Minocyclin + Treatment As Usual (TAU); High Sensitive C-reactive Protein (hs-CRP) > 3mg/L: Minocyclin + Treatment As Usual (TAU)
Drug: Placebo — Oral capsule, no active substance, twice daily, for 12 weeks
  Arms: High Sensitive C-reactive Protein (hs-CRP) < 3mg/L: Placebo + Treatment As Usual (TAU); High Sensitive C-reactive Protein (hs-CRP) > 3mg/L: Placebo + Treatment As Usual (TAU)

SUMMARY:
This is a randomised, double-blind, placebo-controlled clinical trial in which patients with major depressive disorder will receive augmentation through minocycline (MCO), celecoxib (CXB) or placebo.

DETAILED DESCRIPTION:
This project aims to repurpose two established anti-inflammatory compounds as adjuvant therapy for immune-mediated depression, in line with state-of-the-art research of the last 10 years. Immune-mediated depression represents a subtype which accounts for approximately 30% of depressive disorders. Patients with this immunosubtype are more likely to have a higher severity of depression, a lower quality of life and more somatic symptoms. Furthermore it is accompanied by a high incidence of treatment resistance. While their mechanisms of action completely differ from those of existing antidepressant treatment options, immunomodulatory drugs celecoxib and minocycline have proven their merit as add-on treatment in depressive episodes. They have been on the Belgian market for years and come with a known pharmacological and safety profile. Patient stratification at baseline based on inflammatory status will reveal which inflammatory subpopulation benefits most from each of the two investigated anti-inflammatory compounds. Additionally, our distinctive study design allows head-to-head comparison of both add-on therapies and will as such provide the last stepping stones towards clinical implementation of individualised treatment strategies in depression.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 years inclusive.
* Able and willing to give informed consent and take oral medication.
* Physically healthy.
* Diagnosis of Major Depressive Disorder by DSM-5 criteria, confirmed by the Mini International Neuropsychiatric Interview (MINI).
* The current episode of depression has failed to remit to the current antidepressant treatment at the adequate dose (as defined in the Maudsley Prescribing guidelines). Relapse while taking an antidepressant is also considered a treatment failure.
* Tolerant to the current antidepressant and having no planned changes in their current therapy for the duration of the study.
* Stable on current treatment for a minimum of 4 weeks (6 weeks for fluoxetine) prior to baseline.
* If female and of childbearing age, willing to use adequate contraceptive precautions and willing to take a pregnancy test at baseline.

Exclusion Criteria:

* Primary diagnosis of a bipolar disorder, psychotic spectrum disorder, obsessive-compulsive disorder, eating disorder, post-traumatic stress disorder, or alcohol and/or substance use disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (< 4 weeks before screening, excl. nicotine and caffeine).
* Use of immunosuppressant or immunostimulant drugs within 21 days of screening (e.g., glucocorticoid treatment, methotrexate, etc.).
* History of peptic ulcer disease or gastrointestinal (GI) bleeding.
* Having an acute infection or inflammatory bowel disorder.
* Current severe cardiovascular disease, congestive heart failure (NYHA-class II-IV), ischemic or thrombotic events or unstable coronary artery (incl. coronary artery bypass graft (CABG) surgery),
* Liver impairment (alanine aminotransferase > 2x upper limit, serum albumin < 25 g/l or Child-Pugh Score ≥ 10)
* Renal impairment (creatinine clearance < 30 mL/min).
* Having received >14 days of tetracycline or non-steroidal anti-inflammatory medication within the previous 2 months, or having a history of sensitivity or intolerance to these classes of drugs.
* Chronic severe hypertension (systolic BP > 170 mmHg).
* Serology positive for hepatitis-B surface antigen, hepatitis-C antibodies or HIV antibodies.
* Received electroconvulsive therapy < 2 months prior to screening.
* Blood donation in 30 days prior to screening.
* Pregnancy or breastfeeding.
* Currently enrolled in an intervention study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptom severity (HDRS-17) | T0 -> T6 (12 weeks)
  Change in severity of depression measured as the change in the 17-point scale of the Hamilton Depression Rating Scale (HDRS-17; score is ranging from 0 to 52, higher scores indicate higher severity of depressive symptoms) between baseline and endpoint
Remission rate of depression (HDRS-17) | T0 -> T6 (12 weeks)
  Rates of remission measured as a score of ≤7 on the 17-point scale of the Hamilton Depression Rating Scale (HDRS-17; score is ranging from 0 to 52, higher scores indicate higher severity of depressive symptoms and scores 0-7 are considered as being normal) at endpoint

SECONDARY OUTCOMES:
Change in depressive symptom severity (IDS-30SR) | T0 -> T6 (12 weeks)
  Change in severity of depression measured as the change in the Inventory of Depressive Symptomatology - Self Report (IDS-SR; score is ranging from 0 to 84, higher scores indicate higher severity of depressive symptoms)
Response rate of depressive symptoms (HDRS-17) | T0 -> T6 (12 weeks)
  Response rates of the depressive symptoms measured on the 17-point scale of the Hamilton Depression Rating Scale (HDRS-17; score is ranging from 0 to 52, higher scores indicate higher severity of depressive symptoms), with response being defined as a 50% reduction in HDRS-17-score from baseline and partial response as a 25% reduction.
Change in night-time sleep (PSQI) | T0 -> T6 (12 weeks)
  Change in night-time sleep quality and/or quantity measured on the Pittsburgh Sleep Quality Index (PSQI; score is ranging from 0 to 21, higher scores indicate more sleep disturbances)
Change in anxiety (STAI) | T0 -> T6 (12 weeks)
  Change in anxiety measured on the Stait Trait Anxiety Inventory-Self Report (STAI; score is ranging from 20 tot 80, higher scores indicate higher levels of anxiety intensity)
Change in core assessment of psychomotor change (CORE) | T0 -> T6 (12 weeks)
  Change in the degree of psychomotor disturbance (which is as an integral component of melancholia) measured on the Core Assessment Of Psychomotor Change (CORE; score is ranging from 0-54, higher scores indicate higher levels of psychomotor disturbances)
Depressive symptom profiles (IDS-SR) | T0 -> T6 (12 weeks)
  Profile of the depression measured on the Inventory of Depressive Symptomatology - Self Report (IDS-SR; score is ranging from 0 to 84, higher scores indicate higher severity of depressive symptoms)
Therapy compliance (MARS) | T0 -> T6 (12 weeks)
  Therapy compliance measured on the Medication Adherence Scale (MARS; score is ranging from 0-10, higher scores indicate better medication adherence)
Adverse effects | T0 -> T6 (12 weeks)
  Side effects measured with a questionnaire based on the list as used in the Antidepressant Side-Effect Checklist (ASEC-21) and the known side effects of Minocycline and Celecoxib
Metabolic blood markers | T0 -> T6 (12 weeks)
  Cholesterol (mg/dl), High Density Lipoprotein (HDL) (mg/dl), Low Density Lipoprotein (LDL) (mg/dl), fasting glucose (mg/dl), triglycerides (mg/dl)
Other metabolic measures | T0 -> T6 (12 weeks)
  Waist circumference (cm), height (cm) will be measured to calculate the BMI (kg/m^2)
Other metabolic measures | T0 -> T6 (12 weeks)
  Weight (kg) will be measured to calculate the BMI (kg/m^2)

OTHER OUTCOMES:
Immune markers | T0 -> T6 (12 weeks)
  Cytokines: interleukin-6, interleukin-1β, tumor necrosis factor α, interferon γ, Interleukin-1 receptor, interleukin-7
Alternate immune markers | T0 -> T6 (12 weeks)
  Peripheral blood monocytes (PBMCs)
Tryptophan pathway metabolites | T0 -> T6 (12 weeks)
  Kynurenine (KYN), Kynurenic Acid (KYNA), Quinolinic Acid (QA), 3-Hydroxykynurenine (3-HK)
Vascular and (neuro)trophic factors | T0 -> T6 (12 weeks)
  Vascular endothelial growth factor (VEGF), Brain-derived neurotrophic factor (BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Morrens, MD PhD, Principal Investigator — Professor
Locations (3):
- Belgium (3):
  - UPC Duffel, Duffel, Antwerpen
  - UZ Brussel, Brussels
  - Katholiek Universiteit Leuven Campus Kortenberg, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osimo EF, Baxter LJ, Lewis G, Jones PB, Khandaker GM. Prevalence of low-grade inflammation in depression: a systematic review and meta-analysis of CRP levels. Psychol Med. 2019 Sep;49(12):1958-1970. doi: 10.1017/S0033291719001454. Epub 2019 Jul 1. PMID 31258105
- [Background] Foley EM, Parkinson JT, Kappelmann N, Khandaker GM. Clinical phenotypes of depressed patients with evidence of inflammation and somatic symptoms. Compr Psychoneuroendocrinol. 2021 Aug 5;8:100079. doi: 10.1016/j.cpnec.2021.100079. eCollection 2021 Nov. PMID 34729541
- [Background] Carvalho LA, Torre JP, Papadopoulos AS, Poon L, Juruena MF, Markopoulou K, Cleare AJ, Pariante CM. Lack of clinical therapeutic benefit of antidepressants is associated overall activation of the inflammatory system. J Affect Disord. 2013 May 15;148(1):136-40. doi: 10.1016/j.jad.2012.10.036. Epub 2012 Nov 27. PMID 23200297
- [Derived] Wessa C, Janssens J, Coppens V, El Abdellati K, Vergaelen E, van den Ameele S, Baeken C, Zeeuws D, Milaneschi Y, Lamers F, Penninx B, Claes S, Morrens M, De Picker L. Efficacy of inflammation-based stratification for add-on celecoxib or minocycline in major depressive disorder: Protocol of the INSTA-MD double-blind placebo-controlled randomised clinical trial. Brain Behav Immun Health. 2024 Sep 19;41:100871. doi: 10.1016/j.bbih.2024.100871. eCollection 2024 Nov. PMID 39350954